CLINICAL TRIAL: NCT05487612
Title: Minimally Invasive Extracorporeal Circulation Versus Conventional Cardiopulmonary Bypass in Patients Undergoing Cardiac Surgery (MiECS): a Randomised Controlled Trial
Brief Title: MiECC Versus Conventional Cardiopulmonary Bypass in Cardiac Surgery (MiECS)
Acronym: MiECS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Minimal Invasive Extracorporeal Technologies International Society (MiECTiS) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MiECS
Record Dates: First submitted 2022-08-01; First posted 2022-08-04 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Coronary Artery Disease; Aortic Valve Stenosis; Extracorporeal Circulation; Complications
Keywords: Cardiopulmonary bypass; Extracorporeal circulation; Minimal invasive extracorporeal circulation; Coronary artery bypass grafting; Aortic valve replacement
MeSH Terms: conditions — Coronary Artery Disease; Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: Patients undergoing elective or urgent coronary artery bypass grafting, aortic valve replacement or both procedures CABG+AVR using extracorporeal circulation without circulatory arrest will be randomised (1:1 ratio) to having surgery using Minimal Invasive Extracorporeal Circulation (MiECC) or conventional cardiopulmonary bypass (cCPB).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimal Invasive Extracorporeal Circulation (MiECC) (Active Comparator): Patients undergoing coronary artery bypass grafting (CABG), aortic valve replacement (AVR), or combined procedure (AVR+CABG) with Minimal Invasive Extracorporeal Circulation (MiECC).
  Interventions: Device: Minimal Invasive Extracorporeal Circulation
- Conventional Cardiopulmonary Bypass (cCPB) (Active Comparator): Patients undergoing coronary artery bypass grafting (CABG), aortic valve replacement (AVR), or combined procedure (AVR+CABG) with conventional cardiopulmonary bypass (cCPB)
  Interventions: Device: Conventional cardiopulmonary bypass

INTERVENTIONS:
Device: Minimal Invasive Extracorporeal Circulation — Cardiac surgery with Minimal Invasive Extracorporeal Circulation (MiECC).
  Arms: Minimal Invasive Extracorporeal Circulation (MiECC)
Device: Conventional cardiopulmonary bypass — Cardiac surgery with conventional cardiopulmonary bypass (cCPB).
  Arms: Conventional Cardiopulmonary Bypass (cCPB)

SUMMARY:
MiECS is one of the largest multicentre randomised controlled trials on extracorporeal circulation conducted under the auspices of Minimal Invasive Extracorporeal Technologies International Society (MiECTiS). It is designed to ultimately address the emerging effectiveness of MiECC systems in the light of modern perfusion practice worldwide. The primary hypothesis is that MiECC, as compared to conventional CPB (cCPB), reduces the proportion of patients experiencing serious perfusion-related postoperative morbidity after cardiac surgery. The study will be led by the Clinical Research Unit of the Special Unit for Biomedical Research and Education (SUBRE), Aristotle University of Thessaloniki School of Medicine in Greece (AUSoM) with Chief Investigator Professor Kyriakos Anastasiadis, who is a key-opinion-leader in the field of MiECC, founder and Executive Board of MiECTiS.

DETAILED DESCRIPTION:
Despite a fall in mortality rates over the past decade, patients having cardiac surgery continue to experience serious postoperative complications. The risk of serious and relatively common surgical complications is often a consequence of stopping the heart during the operation, using the heart and lung machine (conventional cardiopulmonary bypass; cCPB), and restarting and reperfusing the heart at the end of the operation. Although several strategies have been developed to reduce such complications, they still occur and can be life threatening; they also increase the length of time a patient spends in the hospital.

Miniaturised heart lung machines (minimally invasive extracorporeal circulation; MiECC) have been developed with the aim of reducing the number of postoperative complications arising from using cCPB. Because of the variety of miniaturised systems that have been evaluated, the different types of patients and outcomes investigated, and the poor quality of previous studies, the effectiveness of MiECC in reducing postoperative complications has not been established and most hospitals continue to use cCPB.

Our primary hypothesis is that, compared to cCPB, using a MiECC system during cardiac surgery reduces the proportion of patients having one of several serious postoperative complications (death, myocardial infarction, stroke, acute kidney injury, reintubation, tracheostomy, mechanical ventilation for more than 48 hours, or reoperation) up to 30 days after surgery. In addition, the investigators hypothesise that MiECC reduces the amount of blood products transfused, time to discharge from the cardiac intensive care unit and hospital and the health care resources used during the hospital stay.

Study investigators propose to carry out a large, multicentre randomised controlled trial in 10 to 15 cardiac surgery centres worldwide. Patients will be eligible if they are having coronary artery bypass surgery, aortic valve replace or both using a heart lung machine without circulatory arrest. Centres may recruit patients having all, or a subset of, operation types.

It is expected that 20 % to 23% of patients will experience one or more of the serious complications (the primary outcome). In order to be able confidently to detect a 30% relative reduction in the risk of this outcome, the investigators plan to recruit 1,300 participants across all sites.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing any elective or urgent coronary artery bypass grafting (CABG), aortic valve replacement (AVR) or CABG+AVR surgery using extracorporeal circulation without circulatory arrest.

Exclusion Criteria:

* Requirement for emergency or salvage operation.
* Requirement for major aortic surgery (e.g. aortic root replacement).
* Contraindication or objection (e.g. Jehovah's Witnesses) to transfusion of blood products.
* Congenital or acquired platelet, red cell or clotting disorders (patients with iron deficient anaemia will not be excluded).
* Inability to give informed consent for the study (e.g. learning or language difficulties).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2022-05-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Composite outcome of postoperative serious adverse events | 30 days after randomization following the index admission
  Incidence of: death, postoperative myocardial infarction according to Fourth Universal Definition of myocardial infarction, stroke, all stage acute kidney injury, as defined with AKI Network criteria, Re-intubation, need for mechanical ventilation for > 48 hours, including multiple episodes when separated by more than 12 hours, reoperation and septicaemia confirmed by positive blood culture.

SECONDARY OUTCOMES:
All-cause mortality | 30 days after randomization following the index admission
  All-cause mortality
New-onset postoperative atrial fibrillation | Through initial hospital admission from surgery to initial discharge from hospital, an average of 1 week.
  Incidence of new-onset postoperative atrial fibrillation
Rate of red blood cells transfusion | 30 days after randomization following the index admission
  Units of red blood cells transfused
Rate of platelet transfusion | 30 days after randomization following the index admission
  Units of platelets transfused
Rate of fresh frozen plasma transfusion | 30 days after randomization following the index admission
  Units of fresh frozen plasma transfused
Rate of cryoprecipitate transfusion | 30 days after randomization following the index admission
  Units of cryoprecipitate transfused
Activated Factor VII administration | 30 days after randomization following the index admission
  Incidence of activated factor VII administration
Fibrinogen administration | 30 days after randomization following the index admission
  Incidence of fibrinogen administration
Prothrombin complex concentrate administration | 30 days after randomization following the index admission
  Incidence of prothrombin complex concentrate administration
Time to discharge from cardiac ICU | Through initial hospital admission from surgery to initial discharge from hospital, an average of 1 week.
  Time to discharge from cardiac ICU
Time to discharge from hospital | Through initial hospital admission from surgery to initial discharge from hospital, an average of 1 week.
  Time to discharge from hospital
Delirium | Up to 5 days postoperatively
  Incidence of postoperative delirium
Health-Related Quality of Life (HRQoL) | 90 days after randomization
  HRQoL assessed with EQ-5D questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kyriakos Anastasiadis, Professor, Study Chair — Aristotle University Of Thessaloniki; Polychronis Antonitsis, Assoc. Prof., Study Director — Aristotle University Of Thessaloniki
Locations (12):
- Perfusion Services University Health Network, Toronto General Hospital, Toronto, Canada
- Germany (3):
  - Department of Cardiac Surgery, Coswig
  - Department of Thoracic and Cardiovascular Surgery, University Medical Centre Goettingen, Göttingen
  - Department of Cardiothoracic and Vascular Surgery, Ulm University Hospital, Ulm
- Cardiothoracic Department AHEPA University Hospital, Thessaloniki, Greece
- Italy (2):
  - Department of Cardiac Surgery GVM Anthea Hospital, Bari
  - Department of Cardiac Surgery GVM Maria Eleonora Hospital, Palermo
- Turkey (Türkiye) (2):
  - Department of Cardiovascular Surgery, Ankara City Hospital, Ankara
  - Department of Cardiovascular Surgery, Izmir Bakırçay University, Faculty of Medicine, Izmir
- United Kingdom (3):
  - Department of Cardiac Surgery, Royal Papworth Hospital, Cambridge
  - Deparment of Cardiac Surgery, Castle Hill Hospital, Hull
  - Department of Cardiothoracic Surgery, Hammersmith Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anastasiadis K, Murkin J, Antonitsis P, Bauer A, Ranucci M, Gygax E, Schaarschmidt J, Fromes Y, Philipp A, Eberle B, Punjabi P, Argiriadou H, Kadner A, Jenni H, Albrecht G, van Boven W, Liebold A, de Somer F, Hausmann H, Deliopoulos A, El-Essawi A, Mazzei V, Biancari F, Fernandez A, Weerwind P, Puehler T, Serrick C, Waanders F, Gunaydin S, Ohri S, Gummert J, Angelini G, Falk V, Carrel T. Use of minimal invasive extracorporeal circulation in cardiac surgery: principles, definitions and potential benefits. A position paper from the Minimal invasive Extra-Corporeal Technologies international Society (MiECTiS). Interact Cardiovasc Thorac Surg. 2016 May;22(5):647-62. doi: 10.1093/icvts/ivv380. Epub 2016 Jan 26. PMID 26819269
- [Background] Anastasiadis K, Antonitsis P, Asteriou C, Deliopoulos A, Argiriadou H. Modular minimally invasive extracorporeal circulation ensures perfusion safety and technical feasibility in cardiac surgery; a systematic review of the literature. Perfusion. 2022 Nov;37(8):852-862. doi: 10.1177/02676591211026514. Epub 2021 Jun 17. PMID 34137323
- [Background] COMICS investigators, The COMICS investigators. Conventional versus minimally invasive extracorporeal circulation in patients undergoing cardiac surgery: protocol for a randomised controlled trial (COMICS). Perfusion. 2021 May;36(4):388-394. doi: 10.1177/0267659120946731. Epub 2020 Aug 12. PMID 32781894
- [Background] Wahba A, Milojevic M, Boer C, De Somer FMJJ, Gudbjartsson T, van den Goor J, Jones TJ, Lomivorotov V, Merkle F, Ranucci M, Kunst G, Puis L; EACTS/EACTA/EBCP Committee Reviewers. 2019 EACTS/EACTA/EBCP guidelines on cardiopulmonary bypass in adult cardiac surgery. Eur J Cardiothorac Surg. 2020 Feb 1;57(2):210-251. doi: 10.1093/ejcts/ezz267. No abstract available. PMID 31576396
- [Background] Ranucci M, Johnson I, Willcox T, Baker RA, Boer C, Baumann A, Justison GA, de Somer F, Exton P, Agarwal S, Parke R, Newland RF, Haumann RG, Buchwald D, Weitzel N, Venkateswaran R, Ambrogi F, Pistuddi V. Goal-directed perfusion to reduce acute kidney injury: A randomized trial. J Thorac Cardiovasc Surg. 2018 Nov;156(5):1918-1927.e2. doi: 10.1016/j.jtcvs.2018.04.045. Epub 2018 Apr 18. PMID 29778331
- [Background] Anastasiadis K, Argiriadou H, Deliopoulos A, Antonitsis P. Minimal invasive extracorporeal circulation (MiECC): the state-of-the-art in perfusion. J Thorac Dis. 2019 Jun;11(Suppl 10):S1507-S1514. doi: 10.21037/jtd.2019.01.66. No abstract available. PMID 31293801
- [Background] Kowalewski M, Pawliszak W, Raffa GM, Malvindi PG, Kowalkowska ME, Zaborowska K, Kowalewski J, Tarelli G, Taggart DP, Anisimowicz L. Safety and efficacy of miniaturized extracorporeal circulation when compared with off-pump and conventional coronary artery bypass grafting: evidence synthesis from a comprehensive Bayesian-framework network meta-analysis of 134 randomized controlled trials involving 22 778 patients. Eur J Cardiothorac Surg. 2016 May;49(5):1428-40. doi: 10.1093/ejcts/ezv387. Epub 2015 Nov 3. PMID 26537755
- [Background] Anastasiadis K, Antonitsis P, Papazisis G, Haidich B, Liebold A, Punjabi P, Gunaydin S, El-Essawi A, Rao V, Serrick C, Condello I, Nasso G, Bozok S, Daylan A, Argiriadou H, Deliopoulos A, Karapanagiotidis G, Ashkanani F, Moorjani N, Cale A, Erdoes G, Bennett M, Starinieri P, Carrel T, Murkin J. Minimally invasive extracorporeal circulation versus conventional cardiopulmonary bypass in patients undergoing cardiac surgery (MiECS): Rationale and design of a multicentre randomised trial. Perfusion. 2025 May;40(4):923-932. doi: 10.1177/02676591241272009. Epub 2024 Aug 1. PMID 39089011
- See also: MiECS Clinical Trial Registry by Dendrite — https://miectis.e-dendrite.com